CLINICAL TRIAL: NCT04413357
Title: Plasma Glucose and Insulin Response in Persons with Type 2 Diabetes Mellitus
Brief Title: Glycemic Response in Persons with Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19.01.US.HCN
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — HLA-DM antigens

STUDY DESIGN:
Intervention Model Description: This will be a randomized crossover design. The subjects will be randomized to one of three interventions on three separate study days, one week apart.
Who Masked: Participant
Masking Description: Site pharmacy will not be blinded to product assignment, study staff and participants will be blinded to product assignment. Product will be provided in unlabeled cups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Balanced Nutritional Drink (Active Comparator): The study interventions contain protein, carbohydrate and fat and are intended for use as Supplemental Nutrition.
  Interventions: Other: Balanced Nutritional Drink
- Balanced Nutritional Drink - DMA (Active Comparator): The study interventions contain protein, carbohydrate and fat and are intended for use as retail Supplemental Nutrition for people living with diabetes.
  Interventions: Other: Diabetes Specific, Balanced Nutritional Drink (DMA)
- Balanced Nutritional Drink - DMB (Active Comparator): The study interventions contain protein, carbohydrate and fat and are intended for use as Supplemental Nutrition for people living with diabetes.
  Interventions: Other: Diabetes Specific, Balanced Nutritional Drink DMB

INTERVENTIONS:
Other: Balanced Nutritional Drink — Drink 1 cup of liquid nutrition product that contains protein, carbohydrate and fat intended for use as Supplemental Nutrition.
  Arms: Balanced Nutritional Drink
Other: Diabetes Specific, Balanced Nutritional Drink (DMA) — Drink 1 cup of liquid nutrition product that contains protein, carbohydrate and fat, designed for people living with diabetes and intended for use as Supplemental Nutrition available in retail setting.
  Arms: Balanced Nutritional Drink - DMA
Other: Diabetes Specific, Balanced Nutritional Drink DMB — Drink 1 cup of liquid nutrition product that contains protein, carbohydrate and fat, designed for people living with diabetes and intended for use as Supplemental Nutrition.
  Arms: Balanced Nutritional Drink - DMB

SUMMARY:
This will be a randomized crossover design with nutrition supplement interventions.

DETAILED DESCRIPTION:
This will be a randomized crossover design with three oral nutrition supplement interventions. The subjects will be randomized to one of three interventions on three separate study days, one week apart.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years
* Type 2 diabetes controlled with diet or diet and metformin (Glucophage)
* Hemoglobin A1C less than 9.0%
* Fasting blood glucose less than 180 mg
* Hematocrit levels within normal limits
* Having obtained his/her informed consent

Exclusion Criteria:

* Abnormal thyroid function
* Creatinine >2.0 mg/dl
* Potassium <3.5 mEq/l
* Gastrointestinal disease: ulcer, gastritis, diarrhea, gastroparesis, vomiting
* Currently unstable diabetes or under treatment for cancer, heart disease, renal disease
* Unable to give informed consent or follow instructions
* Current insulin therapy or insulin therapy within the past month
* Patient who are pregnant
* Allergies to milk, soy or any component of the test product
* Patient who in the investigators assessment cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial
* Patients with anemia

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose curve | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
  Area under the blood glucose curve (AUC 0-240 minutes)

SECONDARY OUTCOMES:
Area under the insulin curves | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
  Area under the insulin curves (AUC 0-240)
Insulinogenic index | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
  Insulinogenic index [Change in Ins30/Change in Glu30]

CONTACTS AND LOCATIONS:
Overall Officials: Krysmaru Araujo Torres, MD, Study Director — Nestle Health Science
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No